CLINICAL TRIAL: NCT01365533
Title: A Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Effect of Roflumilast on Airway Inflammation and Function Following Allergen Challenge in Subjects With Allergic Asthma
Brief Title: A Study to Evaluate the Effect of Roflumilast on Airway Inflammation and Function Following Allergen Challenge in Subjects With Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-034
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Allergic Asthma
Keywords: Airway Inflammation; Roflumilast
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roflumilast (Active Comparator)
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast 500 μg, one tablet once daily, orally
  Arms: Roflumilast
Drug: Placebo — Placebo, one tablet once daily, orally
  Arms: Placebo

SUMMARY:
The study was a double-blind, placebo-controlled, crossover study to evaluate the efficacy of roflumilast on airway inflammation and function in patients with allergen-induced asthma.

Individuals with stable, mild to moderate allergic asthma, with a history of episodic wheeze and shortness of breath, were eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* the patient was an outpatient
* had to have a negative (quantitative) serum pregnancy test for female patients of childbearing potential at Phase 1 Screening (Visit 1), a negative urine pregnancy test for female patients of childbearing potential at Phase 3 Randomization/Treatment Period 1 (Visit 5) and Phase 4 Treatment Period 2/Final Evaluation (Visit 9) prior to double-blind treatment
* had symptoms of asthma for the last 6 months that satisfied the American Thoracic Society (ATS) definition of asthma,i.e. episodic wheezing, coughing, shortness of breath, and chest tightness associated with airflow limitation that was at least partially reversible, either spontaneously, or with medication
* had an unmedicated (no inhaled short-acting bronchodilator for at least 8 hours) FEV1 ≥70 percent of the predicted normal value for age, height, and sex, with a 12 percent downward adjustment applied for individuals of African descent
* positive Methacholine (MCh) inhalation challenge at Pre-Randomization Evaluation Visit 2 [provocative concentration resulting in a 20 percent reduction in FEV1 (MCh PC20FEV1) <16 mg/mL] reflecting AHR
* had a documented allergy to a common aeroallergen (animal, dust mite, mold, and pollen allergens) as confirmed by a recognized skin prick test wheal ≥2 mm in diameter.
* positive allergen-induced early and late airway bronchoconstriction. The EAR was defined by an acute fall in FEV1 ≥20 percent within 2 hours following allergen challenge. The LAR was defined by a fall in FEV1 ≥15 percent between 3 hours and 7 hours following allergen challenge
* the patient was someone from whom the investigator or study personnel would expect conscientious cooperation over the duration of the study
* the patient was able to execute or obtain written informed consent at Visit 1.

Exclusion Criteria:

* current neuropsychiatric condition with or without drug therapy that was judged by the investigator to be clinically significant and/or affect the patient's ability to participate in the clinical study. Such as having a history of Attention Deficit/Hyperactivity Disorder (ADHD) that was considered unstable by the investigator, and if pharmacotherapy was required, i.e. Ritalin®, Adderall®, patient had to be on pharmacotherapy for ≥1 month prior to Visit 1. The pharmacotherapeutic regimen had to remain stable during the conduct of the study
* had a history of learning disabilities or intellectual impairment that in the opinion of the investigator prevented the patient from participating in the study
* impairment of hepatic function including alcohol related liver disease, cirrhosis, or hepatitis, cancer, or any clinically significant hematologic, renal, endocrine (except for controlled diabetes mellitus, post-menopausal symptoms, or hypothyroidism), cardiovascular (particularly coronary artery disease, arrhythmias, hypertension, or congestive heart failure), neurologic (including transient ischemic attack, stroke, seizure disorder, migraine headache), or gastrointestinal disease
* clinically significant abnormalities in physical examination and/or in laboratory test results (including hematology and chemistry panels, urinalysis) as assessed by the investigator. The patient was not allowed to have an abnormality detected on physical or laboratory examination considered to be clinically significant by the investigator and limiting to the study's conduct unless the abnormality was related to underlying asthma
* worsening of asthma (requiring daily use of nebulized Beta2-agonists or any use of long-acting Beta-agonists (LABA), or requiring inpatient hospitalization for asthma control, or requiring emergency room treatment, or requiring systemic corticosteroids for asthma control) or respiratory infection in the 6 weeks preceding the Screening Visit
* use of inhaled (>1 mg beclomethasone dipropionate [BDP]-equivalents/day) or systemic (intramuscular, intravenous, or oral) corticosteroids within 60 days prior to Screening and Pre-Randomization Evaluation visits
* use of nasal or inhaled corticosteroids (≤1 mg BDP-equivalents/day), intraophthalmic corticosteroids, nasal, inhaled, or intraophthalmic cromolyn sodium or nedocromil, leukotriene receptor antagonists (zafirlukast,pranlukast, montelukast), and 5-lipoxygenase inhibitors (zileuton) within 4 weeks prior to Screening and Pre-Randomization Evaluation visits. Topical corticosteroids for dermatologic use were allowed
* use of anti-immunoglobulin E (IgE) therapy or immunosuppressives within 3 months prior to Screening and Pre-Randomization Evaluation visits
* use of any immunotherapy within 3 months prior to Screening and Pre-Randomization Evaluation visits
* use of oral and intra-ophthalmic nonsteroidal anti-inflammatory agents (NSAIDs) was permitted, but not within 48 hours of Pre-Randomization Evaluation spirometry. Aspirin® use was not permitted within 7 days of Pre-Randomization Evaluation spirometry
* theophylline-containing agents of any type, LABA (salmeterol, formoterol), and long-acting anticholinergics (tiotropium) were not permitted within 1 week prior to Screening and Pre-Randomization Evaluation visits. Short-acting inhaled Beta2-agonists and inhaled short-acting anticholinergics could be used intermittently according to individual needs, however, they were to be withheld at least 8 hours before the conduct of any challenge or spirometry
* use of oral, intranasal, intra-ophthalmic anti-histamines within 5 days prior to Screening and Pre-Randomization Evaluation visits
* use of caffeine-containing products (such as chocolate, tea, caffeinated sodas) or medications (such as combination products with caffeine, including butalbitalcodeineacetominophen-caffeine, butalbital-acetominophen-caffeine, dihydocodeineacetominophen-caffeine, ergotamine-caffeine, hydrocodone-chlorpheniraminephenylephrineacetominophen-caffeine) for 12 hours, or alcohol or over the counter drugs including cold and allergy medications for 48 hours, or inhaled bronchodilators for 8 hours prior to Screening and Pre-Randomization Evaluation MCh and allergen challenges or spirometry
* herbal supplements and nutraceuticals were not permitted. However, vitamins were allowed
* patient was a smoker (including cigarettes, cigars, pipe, chewing tobacco, or cannabis, i.e. hashish, marijuana). Patients were not allowed to have a history of smoking within the past year and a total smoking history of ≥2 pack-years
* lung disease other than mild to moderate asthma
* concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment could interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease
* recent (<1 year) history of alcohol dependency
* unable and/or unlikely to comprehend and/or follow the protocol over the duration of the study
* participation in any other studies involving investigational or marketed products within 30 days prior to entry into the study
* had donated blood or blood products for transfusion during the 1 month prior to initiation of treatment with study drug, and at any time during the study
* surgery of gastrointestinal tract which could interfere with drug absorption (Note: This was not applicable for minor abdominal surgery such as appendectomy or herniorrhaphy)
* other severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with study participation or investigational product administration or could interfere with the interpretation of study results and, in the judgment of the investigator, could make the patient inappropriate for entry into this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change of percent eosinophils in sputum 24 hours after allergen challenge | From baseline until end of treatment up to 9 weeks
  The primary outcome was the effect of roflumilast on allergen-induced airway eosinophilia.
  Two 15 days treatment periods (14 days with treatment and day 15 without treatment) separated by a washout period (approximately 3 to 5 weeks).

SECONDARY OUTCOMES:
To evaluate the allergen-induced Early asthmatic response (EAR) and Late asthmatic response (LAR) in patients with allergic asthma following repeated dosing of roflumilast | From baseline until end of treatment up to 9 weeks
  * Allergen-induced EAR as measured by Forced expiratory volume in 1 second (FEV1) within 2 hours after allergen challenge, between roflumilast and placebo (Area under the curve [AUC] and maximal drop)
  * Allergen-induced LAR as measured by FEV1 in the period beginning 3 hours and ending 7 hours after allergen challenge, between roflumilast and placebo (AUC and maximal drop)
To evaluate the effect of roflumilast on allergen-induced Airway hyperreactivity (AHR) | From baseline until end of treatment up to 9 weeks
  Allergen-induced AHR at 24 hours post-allergen, as measured by the Methacholine provocative concentration resulting in a 20 percent reduction in FEV1 (MCh PC20FEV1) and as Doubling concentration factor (DC) required to achieve a decrease in FEV1 of 20 percent, between roflumilast and placebo

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed investigational site, Québec, Canada

REFERENCES:
- [Derived] Bardin P, Kanniess F, Gauvreau G, Bredenbroker D, Rabe KF. Roflumilast for asthma: Efficacy findings in mechanism of action studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S4-10. doi: 10.1016/j.pupt.2015.08.006. Epub 2015 Aug 19. PMID 26296794
- [Derived] Gauvreau GM, Boulet LP, Schmid-Wirlitsch C, Cote J, Duong M, Killian KJ, Milot J, Deschesnes F, Strinich T, Watson RM, Bredenbroker D, O'Byrne PM. Roflumilast attenuates allergen-induced inflammation in mild asthmatic subjects. Respir Res. 2011 Oct 26;12(1):140. doi: 10.1186/1465-9921-12-140. PMID 22029856
- See also: BY217-M2-034-RDS-2007-06-05.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4476&filename=BY217-M2-034-RDS-2007-06-05.pdf